CLINICAL TRIAL: NCT05260112
Title: Implementation of a Text Message and Multimedia-based Program for Women Newly Diagnosed With Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: Smartphone-based Self-care Education Program for Women With Interstitial Cystitis: Educational Remote IC Aide
Acronym: ERICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: American Urogynecologic Society (Other)
Responsible Party: Principal Investigator, Lily Arya, Chief, Urogynecology and Reconstructive Surgery, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 844895
Record Dates: First submitted 2022-02-09; First posted 2022-03-02 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Cystitis, Interstitial
Keywords: Self-management; Technology; Text message; Multimedia; Pelvic floor physical therapy; Mindfulness; Cognitive behavioral therapy
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ERICA (Experimental): ERICA is a smartphone-based educational program that teaches women newly diagnosed with interstitial cystitis evidence-based strategies to self-manage their symptoms at home. The program is designed to bridge the interval/gap between initial visit where they are diagnosed with interstitial cystitis and follow up visit. Participants received video learning modules via a secure and HIPAA-compliant text messaging system.
  Interventions: Other: ERICA

INTERVENTIONS:
Other: ERICA — Over 6 weeks, participants receive evidence-based video learning modules twice a week via a secure and HIPAA-compliant text messaging platform. These modules include: patient education on interstitial cystitis, bladder training, trial of an elimination diet, pelvic floor physical therapy including at-home myofascial trigger point release, guided mindfulness practice, and cognitive behavioral therapy for chronic pain.
  At the end of each week, participants receive a check-in message. They also have the opportunity to text questions and concerns, which will be answered using an algorithm-based, clinically validated responses.

SUMMARY:
To implement and assess clinical efficacy of a text message and multimedia-based program that (i) remotely delivers first- and second-line American Urological Association (AUA) treatments of IC/BPS; (ii) integrates treatment of biological (neuropathic pain, pelvic floor dysfunction), psychological (symptom-related fear and anxiety) and social (barriers in access to care, limited patient-provider communication) domains of IC/BPS; (iii) uses clinically validated messages to provide guidance and support.

ELIGIBILITY:
Inclusion criteria:

* Women over 18
* AUA (American Urological Association) criteria for IC/BPS of "an unpleasant sensation (pain, pressure, discomfort) perceived to be related to the urinary bladder, associated with lower urinary tract symptoms of more than six weeks duration, in the absence of infection or other identifiable causes"
* Interested in first- or second-line AUA treatment
* Negative urinalysis and culture within two months of enrollment
* English-speaking
* Own a smartphone with text message and video viewing capability

Exclusion Criteria:

* Women currently on third line or higher treatments
* Currently being treated for UTI
* History of voiding dysfunction such as urinary retention or neurogenic bladder
* Recent (<6 months) pelvic surgery/pregnancy
* Prior pelvic malignancy or radiation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hassani D, Flick L, Sangha H, Brown LA, Andy U, Arya L. How do women with interstitial cystitis/bladder pain syndrome make treatment choices? Int Urogynecol J. 2022 Mar;33(3):583-593. doi: 10.1007/s00192-021-04994-6. Epub 2021 Oct 2. PMID 34599672
- [Background] O'Leary MP, Sant GR, Fowler FJ Jr, Whitmore KE, Spolarich-Kroll J. The interstitial cystitis symptom index and problem index. Urology. 1997 May;49(5A Suppl):58-63. doi: 10.1016/s0090-4295(99)80333-1. PMID 9146003
- [Background] Hanno PM, Erickson D, Moldwin R, Faraday MM; American Urological Association. Diagnosis and treatment of interstitial cystitis/bladder pain syndrome: AUA guideline amendment. J Urol. 2015 May;193(5):1545-53. doi: 10.1016/j.juro.2015.01.086. Epub 2015 Jan 23. PMID 25623737
- [Background] Kanter G, Volpe KA, Dunivan GC, Cichowski SB, Jeppson PC, Rogers RG, Komesu YM. Important role of physicians in addressing psychological aspects of interstitial cystitis/bladder pain syndrome (IC/BPS): a qualitative analysis. Int Urogynecol J. 2017 Feb;28(2):249-256. doi: 10.1007/s00192-016-3109-2. Epub 2016 Aug 31. PMID 27581769
- [Background] FitzGerald MP, Payne CK, Lukacz ES, Yang CC, Peters KM, Chai TC, Nickel JC, Hanno PM, Kreder KJ, Burks DA, Mayer R, Kotarinos R, Fortman C, Allen TM, Fraser L, Mason-Cover M, Furey C, Odabachian L, Sanfield A, Chu J, Huestis K, Tata GE, Dugan N, Sheth H, Bewyer K, Anaeme A, Newton K, Featherstone W, Halle-Podell R, Cen L, Landis JR, Propert KJ, Foster HE Jr, Kusek JW, Nyberg LM; Interstitial Cystitis Collaborative Research Network. Randomized multicenter clinical trial of myofascial physical therapy in women with interstitial cystitis/painful bladder syndrome and pelvic floor tenderness. J Urol. 2012 Jun;187(6):2113-8. doi: 10.1016/j.juro.2012.01.123. Epub 2012 Apr 12. PMID 22503015
- [Background] Lusty A, Kavaler E, Zakariasen K, Tolls V, Nickel JC. Treatment effectiveness in interstitial cystitis/bladder pain syndrome: Do patient perceptions align with efficacy-based guidelines? Can Urol Assoc J. 2018 Jan;12(1):E1-E5. doi: 10.5489/cuaj.4505. Epub 2017 Dec 1. PMID 29173267
- [Derived] Kim EK, Brown LA, Hartzell-Leggin D, Andy UU, Harvie CE, Whitmore KE, Newman DK, Hamm RF, Arya LA. Algorithm-Based Mobile Texting Platform for the Self-Management of Interstitial Cystitis/Bladder Pain Syndrome: Pilot Study Evaluating Feasibility, Usability, and Potential Utility. Urol Pract. 2025 Mar;12(2):203-213. doi: 10.1097/UPJ.0000000000000737. Epub 2024 Oct 11. PMID 39392616

RESULTS

PARTICIPANT FLOW:
Groups:
- ERICA: ERICA is a smartphone-based educational program that teaches women newly diagnosed with interstitial cystitis evidence-based strategies to self-manage their symptoms at home. The program is designed to bridge the interval/gap between initial visit where they are diagnosed with interstitial cystitis and follow up visit. Participants received video learning modules via a secure and HIPAA-compliant text messaging system.
  ERICA: Over 6 weeks, participants receive evidence-based video learning modules twice a week via a secure and HIPAA-compliant text messaging platform. These modules include: patient education on interstitial cystitis, bladder training, trial of an elimination diet, pelvic floor physical therapy including at-home myofascial trigger point release, guided mindfulness practice, and cognitive behavioral therapy for chronic pain.
  At the end of each week, participants receive a check-in message. They also have the opportunity to text questions and concerns, which will be answered using an algorithm-based, clinically validated responses.
Period: Overall Study
Arm/Group | ERICA
Started | 52
Completed | 46
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | ERICA
Number analyzed (Participants) | 52
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 41 [30 to 48]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Female | 49
  Sex/Gender: Non-binary | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 45
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 52
BMI [Mean (Inter-Quartile Range); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 23.8 [22.2 to 27.7]
Duration of IC/BPS symptoms in years [Median (Inter-Quartile Range); unit: years] — Duration in years that participant has had Intercystitis/Bladder Pain Syndrome symptoms
  years | 4 [0.5 to 17]
Duration of IC/BPS diagnosis in years [Median (Inter-Quartile Range); unit: years] — Time in years that participant has been diagnosed with Intercystitis/Bladder Pain Syndrome
  years | 2.5 [0.5 to 15]
Post-menopause [Count of Participants; unit: Participants] — Number of post-menopausal participants
  Participants | 9
Prior treatments: Dietary modification [Count of Participants; unit: Participants] — Number of participants previously treated with dietary modification
  Participants | 12
Prior treatment: Pelvic floor physical therapy [Count of Participants; unit: Participants] — Number of participants previously treated with pelvic floor physical therapy
  Participants | 26
Prior treatment: Bladder analgesic [Count of Participants; unit: Participants] — Number of participants previously treated with bladder analgesics such as Phenazopyridine.
  Participants | 34
Prior treatment: Pentosan polysulfate sodium [Count of Participants; unit: Participants] — Number of participants previously treated with penotsan polysulfate sodium
  Participants | 4
Prior treatment: Tricyclic antidepressant [Count of Participants; unit: Participants] — Number of participants previously treated with tricyclic antidepressant (e.g. amitriptyline)
  Participants | 13
Prior treatment: Antihistamine [Count of Participants; unit: Participants] — Number of participants previously treated with antihistimine, e.g. hydroxyzine
  Participants | 18
Prior treatment: Psychotherapy [Count of Participants; unit: Participants] — Number of participants previously treated with psychotherapy
  Participants | 10
Prior treatment: Mindfulness practice [Count of Participants; unit: Participants] — Number of participants previously treated with mindfulness practice
  Participants | 16
Prior treatment: Yoga [Count of Participants; unit: Participants] | 13
Prior treatment: Cannabinoids [Count of Participants; unit: Participants] | 12
Prior treatment: Prescription opioids [Count of Participants; unit: Participants] — Number of participants previously treated with prescription opioids
  Participants | 3
Prior treatment: Bladder instillation [Count of Participants; unit: Participants] — Number of participants previously treated with bladder instillation
  Participants | 4
Prior treatment: Hydrodistention [Count of Participants; unit: Participants] — Number of participants previously treated with hydrodistention
  Participants | 5
Prior treatment: Fulguration of Hunner lesions [Count of Participants; unit: Participants] — Number of participants previously treated with fulguration of Hunner lesions.
  Participants | 2
Concomitant conditions: anxiety disorder [Count of Participants; unit: Participants] | 35
Concomitant conditions: depressive disorder [Count of Participants; unit: Participants] | 17
Concomitant conditions: anorexia [Count of Participants; unit: Participants] | 4
Concomitant conditions: endometriosis [Count of Participants; unit: Participants] | 8
Concomitant conditions: pelvic inflammatory disease [Count of Participants; unit: Participants] | 2
Concomitant conditions: vulvodynia [Count of Participants; unit: Participants] | 8
Concomitant conditions: irritable bowel syndrome [Count of Participants; unit: Participants] | 13
Concomitant conditions: inflammatory bowel disease [Count of Participants; unit: Participants] | 2
Concomitant conditions: migraine [Count of Participants; unit: Participants] | 16
Concomitant conditions: fibromyalgia [Count of Participants; unit: Participants] | 8
Concomitant conditions: chronic low back pain [Count of Participants; unit: Participants] | 12
Tobacco smoking [Count of Participants; unit: Participants] | 5
Alcohol Use [Count of Participants; unit: Participants] | 27
Provider the IC/BPS diagnosis was made by [Count of Participants; unit: Participants]
  Urogynecologist | 30
  Urologist | 18
  Gynecologist | 2
  Primary Care provider | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Self Efficacy Scale
Description: Validated measure of self-efficacy. Minimum 0 - Maximum 60; higher score means a better outcome
Time Frame: Score at baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ERICA
Number analyzed (Participants) | 52
score on a scale | 10 [2 to 18]
Statistical Analysis 1: Comparison: ERICA; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Interstitial Cystitis Symptom Index
Description: Validated measure of IC/BPS symptom severity. Minimum 0 - Maximum 20; higher score means a worse outcome
Time Frame: Score at baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ERICA
Number analyzed (Participants) | 52
score on a scale | -3 [-5 to -1.5]
Statistical Analysis 1: Comparison: ERICA; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Interstitial Cystitis Problem Index
Description: Validated measure of IC/BPS symptoms' impact on quality of life. Minimum 0 - Maximum 16; higher score means a worse outcome
Time Frame: Scores at baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ERICA
Number analyzed (Participants) | 52
score on a scale | -2 [-5.5 to -0.5]
Statistical Analysis 1: Comparison: ERICA; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Hospital Anxiety and Depression Scale - Anxiety Subscale
Description: Validated measure of anxiety level. Minimum 0 - Maximum 21; higher score means a worse outcome
Time Frame: Score at baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ERICA
Number analyzed (Participants) | 52
score on a scale | -2 [-3 to 0]
Statistical Analysis 1: Comparison: ERICA; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Hospital Anxiety and Depression Scale - Depression Subscale
Description: Validated measure of depression level. Minimum 0 - Maximum 21; higher score means a worse outcome
Time Frame: Score at baseline and 6 weeks.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ERICA
Number analyzed (Participants) | 52
score on a scale | 0 [0 to 0]
Statistical Analysis 1: Comparison: ERICA; Test type: Other; p = 0.53, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Brief Health Care Climate Questionnaire
Description: Validated measure patient's perception of quality of and satisfaction with communication and encounter with the health care system. Minimum 6 - Maximum 30; higher score means a better outcome
Time Frame: Score at baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ERICA
Number analyzed (Participants) | 52
score on a scale | 4 [1 to 9]
Statistical Analysis 1: Comparison: ERICA; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: This study tested a smartphone-based self-management education platform for patients with IC/BPS. No pharmaceutical, procedural, or surgical interventions were involved. No laboratory or diagnostic testings were involved. Thus, there was neither serious adverse event nor mortality events.
Arm/Group | ERICA
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT05260112/Prot_000.pdf
  • Informed Consent Form (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT05260112/ICF_001.pdf